CLINICAL TRIAL: NCT06557447
Title: An Exploratory Clinical Investigation Evaluating Microbiological and Immunological Aspects of Peri-implant Crevicular Fluid and Short-term Treatment Outcomes of Two Different Implant Abutment Surfaces in Subjects Since Four to Nine Years
Brief Title: An Exploratory Clinical Investigation Evaluating Two Abutment Surfaces
Acronym: Exploratory
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Studio Ban Mancini Fabbri (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Efontanarosa
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Peri-implant Crevicular Fluid
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Intervention Model Description: Exploratory study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test Group (Other): Subjects treated between 2019 and 2020 with the NobelActive TiUltra implant and On1 Base Xeal abutment on a previous clinical study protocol approaved by Ethics Committee.
  Interventions: Diagnostic Test: Immunological and microbiological sample of peri-implant crevicular fluid; clinical evaluation
- Control Group (Other): Subjects treated in 2017 with NobelActive TiUnite implant and On1 machined abutment on a previous clinical study protocol approaved by Ethics Committee.
  Interventions: Diagnostic Test: Immunological and microbiological sample of peri-implant crevicular fluid; clinical evaluation

INTERVENTIONS:
Diagnostic Test: Immunological and microbiological sample of peri-implant crevicular fluid; clinical evaluation — Immunological sample collection involves placing a Periopaper strip in the peri-implantar sulcus for 30 seconds. If sample is contaminated with blood, sample will be discarded and another sample will be collected (a different surface of the same implant/tooth can be used).
  Microbiological sample collection involves collecting subgingival dental plaque by sliding the end of the STERILE curette (Gracey) inside the peri-implant sulcus. In case of slight bleeding following the first sample, dry the site again before collection. In case of profuse bleeding, collect a sample from another site (by site mean mesial/buccal/distal/lingual) of the same implant.
  Both immunological and microbiological samples will be sent for respective laboratories for the analysis.
  Clinical evaluation will assess presence of dental plaque, bleeding on probing and gingival status.

SUMMARY:
A total of 22 subjects will be included in the study. The subjects who were treated with NobelActive TiUnite and On1 machined abutment will be enrolled in the control group and subjects who were treated with NobelActive TiUltra and On1 Base Xeal abutments will be enrolled in the test group. Two peri-implant crevicular fluid (PICF) samples will be collected for immunological testing and two plaques samples will be collected for microbiological testing from all the enrolled subjects one from the control/test implant site and one from the contralateral tooth/implant site. 3 weeks after the first sampling PICF and plaques sampling will be repeated the same way.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the clinical, microbiological, and immunological biomarkers of implant sites which were treated with two different implant-abutment-systems (anodized surface and machined surface). This single-center exploratory study includes 22 subjects, divided into two distinct groups: Test group and Control group. All subjects in both groups have undergone treatment. In the Test group, subjects were treated between 2019 and 2020 with the NobelActive TiUltra implant and On1 Base Xeal abutment, while in the Control group, treatment occurred in 2017 with NobelActive TiUnite implant and On1 machined abutment. All subjects were treated by the same clinician, Dr Giacomo Fabbri, and were participants in two approved clinical study protocols (T-190 and IIT 2017-1538) approaved by local Ethics Committee. T-190, a multicenter study, involved 21 subjects from Dr Fabbri's center, with 12 subjects available for recall (Control group) in this study. The IIT 2017-1538 study included 61 subjects, with 12 subjects scheduled for recall (Test group) in the current study. Two subjects were part of both the studies, received both the implant abutment solutions and belong to both the groups. The subjects are enrolled provided they meet all the inclusion and none of the exclusion criteria and sign the informed consent. Peri-implant crevicular fluid (PICF) and plaques samples will be collected from control and test implant sites (and respective contralateral tooth/implants) of each participating subject for immunological and microbiological testing at two time points with an interval of approximately 3 weeks between the two sample collections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to sign the Informed Consent Form
* Subjects able to adhere to the investigation schedule
* Subjects with no previous surgical intervention or soft tissue complications in the area of the implant site (e.g., localized mucositis, mild peri-implantitis, etc.) within 3 months before first sample collection
* Subjects regularly adhere to a professional oral hygiene maintenance program
* No recent antibiotics or biological therapy (or any treatment that activates or suppresses the immune system)
* No xerostomia

Exclusion Criteria:

* Subject not willing to sign the Informed Consent Form
* Subject not able to adhere to the investigation schedule

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate immunological markers in peri-implant crevicular fluid | 2 samples collections with 3 weeks of interval
  Immunological sample collection of subgingival area (per-implant crevicular fluid) on implant and contralateral tooth/implant for test and control group
Evaluate microbiological response in peri-implant crevicular fluid | 2 samples collections with 3 weeks of interval
  Microbiological sample collection of subgingival area (per-implant crevicular fluid) on implant and contralateral tooth/implant for test and control group
Bleeding Index | Pre-treatment/initial visit
  Bleeding on probing will be assessed on implant and contralateral tooth/implant for test and control group
Gingival Index | Pre-treatment/initial visit
  Gingival status will be assessed on implant and contralateral tooth/implant for test and control group
Plaque Index | Pre-treatment/initial visit
  Dental plaque will be assessed on implant and contralateral tooth/implant for test and control group

IPD SHARING:
Plan to Share IPD: No